CLINICAL TRIAL: NCT02535130
Title: Evaluation of Nebulization and Positive Expiratory Pressure Combination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NebuPEP
Record Dates: First submitted 2015-08-24; First posted 2015-08-28 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Cystic Fibrosis; Healthy Subjects
MeSH Terms: conditions — Cystic Fibrosis | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebulization combined to positive expiratory pressure (Experimental): Experimental arm
  Interventions: Device: Positive expiratory pressure; Drug: amikacine nebulization
- Nebulization (Active Comparator): Control arm
  Interventions: Drug: amikacine nebulization

INTERVENTIONS:
Device: Positive expiratory pressure
  Arms: Nebulization combined to positive expiratory pressure
Drug: amikacine nebulization

SUMMARY:
The purpose of this study is to compare the efficiency of nebulization and positive expiratory pressure combination

ELIGIBILITY:
Inclusion Criteria:

* Stable cystic fibrosis patients older than 16 y.o.
* Healthy subjects

Exclusion Criteria:

* Kidney failure
* No pregnancy

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Urinary excretion of amikacin | 24 hours after the nebulization
  Pharmacokinetic study of the urinary excretion of amikacin after nebulization

SECONDARY OUTCOMES:
breathing pattern | participants will be recorded for the duration of the nebulization, an expected average of 15 minutes
  recoding of frequency and tidal volume during the nebulization

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Aubriot AS, Leal T, Dubus JC, Gohy S, Reychler G. Impact of adding positive expiratory pressure to nebulisation on drug delivery: a comparative study. Physiotherapy. 2025 Feb 13:101772. doi: 10.1016/j.physio.2025.101772. Online ahead of print. PMID 40199650